CLINICAL TRIAL: NCT04079192
Title: A Prospective, Randomized, Non-Inferiority Trial to Determine the Safety and Efficacy of the BA9TM Drug Coated Balloon for the Treatment of In-Stent Restenosis: First-in-Man Trial (REFORM)
Brief Title: Biolimus A9™ (BA9™) Drug Coated Balloon (DCB) Study
Acronym: REFORM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biosensors Europe SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-EU-01
Record Dates: First submitted 2019-08-27; First posted 2019-09-06 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Coronary Artery Disease; In-Stent Restenosis
Keywords: Drug-Coated Balloon
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients who meet all the eligibility criteria will be randomized 2:1 to receive treatment with either a BA9-DCB or a Sequent Please® Paclitaxel Coated Balloon.
Who Masked: Participant
Masking Description: The subject will be blinded to the study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biolimus A9™ Drug Coated Balloon (Experimental): Patients who meet the eligibility criteria and who are randomised to this arm, will receive treatment with the Biolimus A9™ Drug Coated Balloon
  Interventions: Device: Biolimus A9 Drug Coated Balloon
- Sequent ® Please Paclitaxel coated balloon (Active Comparator): Patients who meet the eligibility criteria and who are randomised to this arm, will receive treatment with the Sequent ® Please Paclitaxel coated balloon
  Interventions: Device: SeQuent Please Paclitaxel Drug Coated Balloon

INTERVENTIONS:
Device: Biolimus A9 Drug Coated Balloon — A non-surgical procedure that uses a catheter to place a semi-compliant angioplasty drug coated balloon to open up coronary arteries that have been narrowed by atherosclerosis. The balloon is inflated to treat the stenosis and transfer the drug to arterial wall, and then is deflated and withdrawn.
  Arms: Biolimus A9™ Drug Coated Balloon
Device: SeQuent Please Paclitaxel Drug Coated Balloon — A non-surgical procedure that uses a catheter to place a semi-compliant angioplasty drug coated balloon to open up coronary arteries that have been narrowed by atherosclerosis. The balloon is inflated to treat the stenosis and transfer the drug to arterial wall, and then is deflated and withdrawn.
  Arms: Sequent ® Please Paclitaxel coated balloon

SUMMARY:
The study is a Prospective, Randomized, Non-Inferiority Trial to Determine the Safety and Efficacy of the BA9™ Drug Coated Balloon for the Treatment of In-Stent Restenosis. It is a First-in-Man Trial.

DETAILED DESCRIPTION:
This clinical trial will serve as a first-in-human (FIH) experience for the BA9™ DCB in a population of patients with coronary artery disease who have an indication for interventional treatment of in-stent restenosis (ISR) in a bare-metal stent (BMS) or drug-eluting stent (DES).

The study uses a prospective, multi-center, single blind, randomized controlled trial design to enroll 195 patients. The study will seek to prove that the BA9-DCB is non-inferior to the approved CE marked Sequent Please® Paclitaxel Coated Balloon with respect to % Diameter Stenosis and has similar safety characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with in-stent restenosis (ISR) and clinical symptoms of ischemia and/or (i) evidence of ischemia on non-invasive testing or (ii) hemodynamically relevant lesion defined by FFR ≤ 0.80 or iFR ≤ 0.89 or > 90% stenosis.
* Patient presenting with a lesion that can be fully covered with one DCB length. - Patients can have up to two index lesions with ISR, which can both be treated and evaluated.
* Patient has provided written informed consent
* Age ≥ 18 years.
* Patient is willing and able to comply with the study procedures and follow-up.

Exclusion Criteria:

* Patient presents with a ST-elevation myocardial infarction (STEMI) or had an acute MI within 48 hours prior to presentation (according to the universal definition of myocardial infarction).
* Patient with acute cardiac decompensation or acute cardiogenic shock
* Documented left ventricular ejection fraction (LVEF) ≤ 30%
* Patient with impaired renal function (glomerular filtration rate < 80 mL/min/1.73 m2).
* More than 2 epicardial vessels requiring revascularization
* Significant left main stenosis (by visual estimation) or an ISR located in the left main (LM).
* Patient has an ISR lesion that cannot be covered with one DCB length.
* Patient has an ISR in the target segment in a stent of a smaller diameter than 2.5mm.
* Severe calcification that might prevent a sufficient expansion of the DCB, if not pre-treated with rotablation or a shockwave application device.
* Known hypersensitivity or contraindication to biolimus, paclitaxcel, aspirin, thienopyridines, or iodinated contrast that cannot be pre-treated.
* Pregnant and/or breast-feeding females or females who intend to become pregnant during the time of the study.
* Subject currently enrolled in other investigational device or drug trial in which the primary endpoint has not yet been reached.
* Anticipated difficulties to complete the angiographic follow-up study.
* Patient with a life expectancy of less than 12 months.
* Patients lacking mental capacity (i.e. patients suffering from dementia and others) to provide informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Percent Diameter Stenosis (DS) | 6 months
  Percent DS of the target segment assessed by quantitative coronary angiography (QCA)

SECONDARY OUTCOMES:
Target lesion failure | 1 month, 6 months, 1 year and 2 years
  Taget lesion failure defined as a composite of cardiovascular death, any target vessel myocardial infarction, coronary artery bypass graft and clinically driven target lesion revascularization
Target vessel failure | 1 month, 6 months, 1 year and 2 years
  Target vessel failure defined as a composite of cardiovascular death, any target vessel myocardial infarction, and clinically driven target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Byrne, MD, PhD, Principal Investigator — Mater Private Hospital
Locations (15):
- Germany (3):
  - Heart Center, Segeberger Kliniken, Bad Segeberg
  - Heart Center Leipzig - University of Leipzig, Leipzig
  - Evangelisches Krankenhaus Paul Gerhardt Stift, Wittenberg
- Ireland (2):
  - Mater Private Hospital, Dublin
  - University Hospital Galway, Galway
- Centro Cardiologico Monzino, Milan, Italy
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de La Princesa, Madrid
- United Kingdom (6):
  - Royal Bournemouth hospital, Bournemouth
  - University Hospital of Wales, Cardiff
  - Craigavon Cardiac Centre, Craigavon
  - Dorset County Hospital, Dorchester
  - Altnagelvin Area Hospital, Londonderry
  - Worcestershire Royal Hospital, Worcester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Byrne RA, Hahn JY, O'Kane P, Sabate M, Toelg R, Copt S, Fitzgerald S, Morice MC, Trevelyan J, Mylotte D, Ortiz AF, Rai H, Durand R, Wohrle J, Kleber FX, Stefanini G, Alfonso F. Randomized Trial of Biolimus DCB for In-Stent Restenosis: The Primary Results of the REFORM Study. JACC Cardiovasc Interv. 2025 Mar 10;18(5):654-662. doi: 10.1016/j.jcin.2024.11.026. Epub 2025 Feb 5. PMID 39918494
- [Derived] Traynor BP, Fitzgerald S, Alfonso F, O'Kane P, Sabate M, Tolg R, Trevelyan J, Hahn JY, Mylotte D, Wohrle J, Rai H, Cortese B, Morice MC, Schuette D, Copt S, Oldroyd KG, Byrne RA; REFORM investigators. Design and rationale of a prospective, randomized, non-inferiority trial to determine the safety and efficacy of the Biolimus A9 drug coated balloon for the treatment of in-stent restenosis: First-in-man trial (REFORM). Cardiovasc Revasc Med. 2023 Nov;56:75-81. doi: 10.1016/j.carrev.2023.06.004. Epub 2023 Jun 6. PMID 37328392